CLINICAL TRIAL: NCT06437028
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Evaluating the Efficacy of Multiple Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus Standard of Care Alone in the Treatment of Nonhealing Diabetic Foot Ulcers.
Brief Title: Evaluating the Efficacy of Perinatal Membrane Allografts in Addition to the Standard of Care for the Treatment of Non-healing Diabetic Foot Ulcers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samaritan Biologics (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SB-24-01
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Diabetic Foot; Allograft; Amnion; Chorion; Wound healing; Advanced wound care; Comparative effectiveness; Lower extremity ulcer; Time to heal; Treatment; Diabetes complication; Skin ulcer; Neuropathy; Peripheral artery disease; Ischemia; Wagner Grade
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Leg Ulcer; Diabetes Complications; Skin Ulcer; Peripheral Arterial Disease; Ischemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study will be modified platform design in which two treatment groups will be compared to one control group initially. However, this study design will enable the inclusion of additional study groups over time while concomitantly increasing the control group size to maintain adequate power.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dual-layer perinatal tissue allograft (Experimental): Patients will receive weekly applications of a dual-layer perinatal tissue allograft in addition to standard of care wound management.
  Interventions: Other: Dual-layer perinatal tissue allograft; Other: Standard of care
- Three-layer fenestrated perinatal tissue allograft (Experimental): Patients will receive weekly applications of a three-layer fenestrated perinatal tissue allograft in addition to standard of care wound management.
  Interventions: Other: Three-layer fenestrated perinatal tissue allograft; Other: Standard of care
- Standard of care (SOC) wound management (Active Comparator): Standard of care (SOC) will include cleansing of the index wound with sterile normal saline solution, followed by sharp debridement to remove necrotic tissue, application of appropriate dressings and wound off-loading.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Dual-layer perinatal tissue allograft — The dual-layer perinatal tissue allograft is an amnion - amnion allograft
  Arms: Dual-layer perinatal tissue allograft
Other: Three-layer fenestrated perinatal tissue allograft — The three-layer fenestrated perinatal tissue allograft is an amnion - chorion - amnion allograft
  Arms: Three-layer fenestrated perinatal tissue allograft
Other: Standard of care — Standard of care (SOC) will include cleansing of the index wound with sterile normal saline solution, followed by sharp debridement to remove necrotic tissue, application of appropriate dressings and wound off-loading.

SUMMARY:
The goal of this clinical trial is to learn if using perinatal tissue allografts improves healing of chronic, non-healing foot ulcers in diabetic patients.

The main question that this study aims to answer is:

Does the use of perinatal tissue allografts in conjunction with standard of care wound management techniques result in a higher percentage of target ulcers achieving complete closure (i.e. healing) as compared to ulcers being treated with standard of care alone after 12 weeks of treatment.

One ulcer on each participant's foot will receive weekly 1) applications of perinatal tissue allografts and standard of care wound management or 2) standard of care wound management alone. Pictures of the ulcer and measurements of its size will be measured every week to track its healing progress over a total treatment period of 12 weeks. Additionally, the participants will be asked to fill out a questionnaire about the wound impacts their life and their quality of life.

DETAILED DESCRIPTION:
Patients with diabetes often develop ulcers on their lower extremities. While some ulcers can be managed using standard of care wound management techniques including debridement, moist dressings, infection control and off-loading, many develop into chronic, non-healing wounds. Chronic non-healing wounds can lead to higher risk of infection, amputation and decreased quality of life.

Advanced wound therapies aim to promote rapid and complete healing of chronic wounds. An example of an advanced wound therapy are perinatal tissue allografts. These include human amniotic / chorionic membranes, which have been confirmed by the United States Food & Drug Administration's Tissue Reference Group to meet the criteria for regulation solely under Section 361 of the Public Health Service Act as defined in Title 21 of the Code of Federal Regulations - Part 1271 for the management of diabetic foot ulcers.

The focus of this clinical trial is to determine the clinical utility of treating diabetic foot ulcers with weekly applications of perinatal tissue allografts in addition to standard of care wound management techniques compared to applying standard of care wound management only.

It is hypothesized that the addition of perinatal tissue allografts to standard of care treatment will result in a higher percentage of ulcers achieving complete closure (i.e. healing) compared to ulcer being treated with standard of care alone after 12 weeks of treatment.

To test this hypothesis the study will consist of patients who will undergo a 2-week screening phase and a 12-week treatment phase. Briefly, during the 2-week screening phase, patients meeting inclusion criteria will have an identified index wound managed with standard of care. Index wounds that are not reduced by more than 20% in the screening phase will be randomized into the treatment groups. During the 12-week treatment phase, index wounds will be treated weekly with either allograft and standard of care or standard of care alone.

Evaluation of data (outcome measures) associated with the trial will include intent to treat and per protocol analyses which will be performed by at least one blinded statistician and investigator.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are required to meet all the following criteria for enrollment in the study.

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment in the study.

1. A subject known to have a life expectancy of < 6 months is excluded.
2. The subject is excluded if the target ulcer is not secondary to diabetes.
3. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
4. If there is evidence of osteomyelitis complicating the target ulcer, the subject is excluded.
5. A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
6. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
7. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
8. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
9. The subject is excluded if the surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Photographic planimetry is not required for measurements taken during the historical run-in period (e.g. calculating surface area using length x width is acceptable).
10. The subject is excluded if the surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1/randomization visit, during which time the subject received SOC.
11. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
12. A subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
13. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
14. A potential subject with end stage renal disease requiring dialysis is excluded.
15. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
16. A subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
17. A Subject treated with hyperbaric oxygen therapy or a Cellular Acellular, or Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit is excluded.
18. A subject is excluded if they are malnourished: a score of less than 17 on the Mini Nutritional Assessment (MNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complete Wound Closure | 12-weeks following study screening phase
  The percentage of wounds completely healed. Complete healing will be defined as 100% epithelialization without drainage and need for dressing or wound size ≤ 0.1cm^2 as determined by the site investigator and validated by a blinded review board.

SECONDARY OUTCOMES:
Time to wound closure | 12-weeks following study screening phase
  Time to wound closure over 12 weeks will be determined via a Kaplan-Meier analysis
Percent reduction in wound area | 12-weeks following study screening phase
  Percent reduction of wound area [(Ai-Axw]) / Ai] x100, where Ai is the area of the index wound at randomization, Axw is the wound area at weekly intervals.
Reduction in Adverse Events | 12-weeks following study screening phase
  A symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries will be regarded as adverse events. Abnormal results of laboratory or diagnostic procedures are considered to be adverse events if the abnormality:
  1. Results in study withdrawal.
  2. Is associated with a serious adverse event.
  3. Is associated with clinical signs or symptoms.
  4. Leads to additional treatment or to further diagnostic tests.
  5. Is considered by the Investigator to be of clinical significance
Forgotten Wound Score Measure | 12-weeks following study screening phase
  Forgotten Wound Score Measure
Wound Quality of life questionnaire | 12-weeks following study screening phase
  Wound-QoL questionnaire on quality of life with chronic wounds

OTHER OUTCOMES:
Proportion of ulcers that completely heal in patients 65 years or older | 12-weeks following study screening phase
  Proportion of ulcers that completely heal in patients 65 years or older for CAMP plus SOC versus SOC alone

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- Monroe Biomedical Research, Monroe, North Carolina, United States